CLINICAL TRIAL: NCT00005105
Title: Genetic Study of Insulin-Like Growth Factor-I Receptor Mutations in Patients With Intrauterine Growth Retardation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Other Study IDs: 199/14924; CHMC-C-96-10-4
Record Dates: First submitted 2000-04-06; First posted 2000-04-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Intrauterine Growth Retardation
Keywords: endocrine disorders; intrauterine growth retardation; rare disease
MeSH Terms: conditions — Fetal Growth Retardation; Endocrine System Diseases; Rare Diseases

SUMMARY:
OBJECTIVES:

I. Determine if mutations in the gene encoding the insulin-like growth factor-I receptor lead to relative insulin-like growth factor-I insensitivity and produce intrauterine growth retardation in children.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients undergo blood draw. Insulin-like growth factor-I (IGF-I) and insulin-like growth factor binding protein-3 (IGFBP-3) are measured. Patients whose IGF-I and IGFBP-3 levels are average or above are tested for the presence of mutation in the insulin-like growth factor-I receptor.

ELIGIBILITY:
* Intrauterine growth retardation (IUGR), defined as birth weight less than 2 standard deviations below the mean by Usher and McLean Deficient "catch-up" growth (stature less than 5th percentile on growth chart after age 18 months) Normal or elevated circulating concentrations of insulin-like growth factor-I (IGF-I) and insulin-like growth factor binding protein-3 (IGFBP-3) IGF-I or IGFBP-3 within or above the 95th percentile confidence interval for age No other clinical explanation for poor prenatal and postnatal growth No IUGR due to maternal toxemia, endocrine disease, gastrointestinal disease, significant heart disease, or chromosomal abnormalities No other condition known to retard growth

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75
Dates: Start 1997-01

CONTACTS AND LOCATIONS:
Overall Officials: Steven D. Chernausek, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - Emory University School of Medicine, Atlanta, Georgia
  - James Whitcomb Riley Hospital for Children, Indianapolis, Indiana
  - Schneider Children's Hospital, New Hyde Park, New York
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Medical College of Virginia School of Medicine, Richmond, Virginia